CLINICAL TRIAL: NCT03348007
Title: A Randomized Double-blind Placebo-controlled Clinical Trial Assessing the Efficacy and Safety of Hépar® in Chronic Constipation
Brief Title: Clinical Trial Assessing the Efficacy and Safety of Hépar® in Chronic Constipation
Acronym: HEP02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-A00948-39
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized (2-arm), double-blind, comparative study versus weakly mineralized water (placebo) in women with functional constipation (Rome Criteria III).
  During the selection visit functional constipation will be evaluated by retrospective examination over the previous 3 months according to the diagnostic criteria for functional constipation in Rome III. During the 7 to 9 days prior to randomization, the patients selected by the investigators will observe a period of Wash out and will have to drink 1.5l of Nestlé PureLife® (low mineral water) water per day and inform them daily about their symptomatology ( stool frequency, abdominal pain aspect), their water intake and rescue laxative treatment.
  Wash-out period concerned previous taking of laxatif drugs
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEPAR (Experimental): 1L of Hépar + 0.5L of low-mineral water (Hépar group).
  Interventions: Other: Taking two kinds of mineral water
- VITTEL Bonne Source (Active Comparator): 1.5L of low-mineral water (Vittel Bonne Source, control group)
  Interventions: Other: Taking two kinds of mineral water

INTERVENTIONS:
Other: Taking two kinds of mineral water — 1.5L of low-mineral water (Vittel Bonne Source, control group) or 1L of Hépar + 0.5L of low-mineral water (Hépar group).

SUMMARY:
The study objectives are to evaluate the efficacy and safety of a 2-week daily intake of 1L Hépar® natural mineral water rich in magnesium sulphate compared to a control natural mineral water in the treatment of the constipation symptoms in women outpatients.

DETAILED DESCRIPTION:
Healthy patients meeting all of the following criteria were included in the study: i) female outpatient aged 18 to 60, ii) with a diagnosis of functional constipation according to the Rome III criteria for 3 months or more, iii) without any laxative drug for 3 days prior to inclusion, iv) having easy access to toilet, v) regularly eating vegetables and fruits, vi) having physical activity, reasonable walking periods or exercise 2 or 3 times a week and vii) drinking 1.5±0.5L of water /day. Patients who presented any of the following criteria were excluded from the study: i) known unsatisfaction to Hépar, ii) concomitant treatment or disease (current or past) likely to interfere with evaluation of the study parameters and iii) documented pregnancy. The study was conducted by 28 city-based general practitioners located throughout France.

After a screening visit, patients followed a washout during 7 to 9 days before inclusion. Patients had to stop any drug treatment liable to interfere with transit and drink 1.5 litres per day of a low-mineral spring water (Nestlé Purelife, Nestlé Waters, France). At the inclusion visit, patients were randomized to the control or Hépar group according to the chronological order of inclusion and to a predetermined randomization list in balanced blocks of 4 treatment units (SAS® software). The randomization list was prepared in advance by the statistician from the society in charge of the logistic of bottles, and secured in an electronic file with restricted access. Two sets of sealed envelopes kept by the investigator and the study manager in a secure and locked place were generated to contain the patient's randomization number and allocated group. The investigator could break the blinding in case of absolute emergency and in accordance with the sponsor. The follow-up visit was performed 15 to 17 days following inclusion.

Patients had to drink 1.5L per day from day 1 to day 14. Depending of the randomization, they drank either 1.5L of low-mineral water (Vittel Bonne Source, control group) or 1L of Hépar + 0.5L of low-mineral water (Hépar group).

During the screening visit (V0), the physician collected sociodemographics, previous medical history and history of the constipation episode (Rome III criteria), onset of symptoms, abdominal pain on a 100 mm VAS, dietary habits, physical activities and previous and current treatments. The patient was provided with a self-evaluation e-diary to collect: i) the number and type of stools (Bristol Scale); ii) abdominal pain, iii) physical activity and iv) drug, water, beverage and food consumption during washout.

At inclusion (V1), the physician collected: i) the weekly number and type of stools, ii) Rome III criteria, iii) AEs, iv) ability to complete the e-diary, v) compliance to the washout treatment (count of unused bottles), and vi) use of rescue medication over the past week.

During the final visit (V2), the physician collected: i) the weekly number and type of stools, ii) Rome III criteria, iii) AEs, iv) compliance to the treatment (count of unused bottles) and v) use of rescue medication over the past two weeks.

For the washout and the treatment periods, the type of stools was assessed directly by the patient on the e-diary and secondarily by an independent expert, based on the photographs the patient had to make of each of their stools.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 18 to 60.
* Outpatients.
* Diagnosis of constipation according to the Rome III criteria Symptoms ≥3 months Onset ≥6 months prior to diagnosis

  a. Presence of ≥2 of the following symptoms for at least 25% of defecations: straining, lumpy or hard stools, sensation of incomplete evacuation, sensation of ano-rectal obstruction/blockage, manual maneuvers to facilitate defecation (e.g., digital evacuation, support of the pelvic floor), <3 defecations/week and b. Loose stool rarely present without use of laxative and c. Insufficient criteria for Inflammatory Bowel Syndrome with constipation (IBS-C)
* No laxative drug for ≥ 3 days preceding the inclusion.
* Easy access to toilet at work or elsewhere.
* Regularly consumption of vegetables and fruits.
* Physical activity 2 or 3 times a week.
* Consumption of 1.0 L to 1.5 L of water per day.
* Signed informed consent.
* Ability to follow the study instructions.
* Health insurance coverage.

Exclusion Criteria:

* Current pregnancy.
* Severe or acute disease likely to interfere with the results of the study or to be life-threatening.
* History of digestive disease, digestive malformation.
* Metabolic disease.
* Dysfunction of phospho-calcium metabolism.
* History of renal disease (renal insufficiency etc.) or cardio-vascular disease (cardiac insufficiency...), respiratory disease, neural disease.
* Subject on local or general treatment (prescribed drugs, food supplements etc.) likely to interfere with evaluation of the study parameters, including hydration status and transit.
* Subject who refuses to sign the declaration of informed consent.
* Subject not available for the entire duration of the study.
* Subject having a bad acceptance to Hépar® water.
* Subject being currently treated with drugs that can interact on digestive motility: paraffin, mucilages, pro or prebiotics, lactulose, lactitol, PEG.
* Subject has participated in a clinical trial within 3 months prior to baseline visit.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 262 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2016-07-22 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal transit | day 14
  The primary study endpoint will be the gastro-intestinal transit change measured by the percentage of responder subjects defined as a composite score of the two following Rome III criteria:
  number of stools ≥ 4 or an increase of 2 stools/week and stools consistency with less than 25% of lumpy to hard stools reviewed by an independent expert on objectified criteria (photography)

SECONDARY OUTCOMES:
Defecation frequency | day 14
  frequency questionnaire
Stool consistency | day 14
  Bristol stool scale The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories. It is used in both clinical and experimental fields.
  The seven types of stool are:
  Type 1: Separate hard lumps, like nuts (hard to pass); also known as goat faeces Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid
Intensity/severity of the patient's constipation | day 14
  based on the global score and on each of the 17-items of the Rome III constipation module questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Baudouin TCHAKONTE, MD, Principal Investigator — 44340 Bouguenais France
Locations (1):
- Quanta Medical, Rueil-Malmaison, France

IPD SHARING:
Plan to Share IPD: No